CLINICAL TRIAL: NCT05918146
Title: Effects of Hypertonic Dextrose Prolotherapy on Conventional Physical Therapy in Patients With Subdeltoid Bursitis: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Dextrose Therapy on Physical Therapy in Subdeltoid Bursitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023SKHADR033
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Subdeltoid Bursitis; Injection; Effect of Drug
Keywords: subdeltoid bursitis; dextrose; physical therapy
MeSH Terms: interventions — Glucose; Physical Therapy Modalities; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dextrose injection, one time
  Interventions: Drug: Dextrose
- Control group (Placebo Comparator): Normal saline injection, one time
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dextrose — Dextrose injection plus physical therapy
  Other Names: physical therapy
  Arms: Intervention group
Drug: Normal saline — Normal saline injection plus physical therapy
  Other Names: physical therapy
  Arms: Control group

SUMMARY:
Physical therapy and hypertonic dextrose prolotherapy are often used to treat subdeltoid bursitis. This study aims to investigate the effects of hypertonic dextrose injection on physical therapy through a double-blind, randomized study.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled clinical trial will be conducted to collect 44 patients with subdeltoid bursitis. In the first week and the third week, a total of 20% hypertonic dextrose 10 mL (experimental group) and normal saline 10 mL (placebo group) will be injected under sonographic guidance, and physical therapy (hot shoulder pack, interference wave, and exercise for 20 minutes each) 3 times per week for one month will be arranged. Shoulder pain by visual analog scale, function (including Disabilities of the Arm, Shoulder, and Hand: DASH and Shoulder Pain and Disability Index: SPADI), quality of life (Brief version of the World Health Organization Quality of Life Scale: WHOQOL-BREF) and high-resolution ultrasound examination will be arranged at before treatment, one week after treatment (i.e., one week after injection), one month, and three months after injection.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of subdeltoid bursitis age 20 or older 20 at least one positive in the painful arc, neer test, or Hawkins test can attend 3 months of intervention and follow up

Exclusion Criteria:

* history of malignancy previous shoulder operation or injury previous shoulder injections in the past 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder pain and disability, ranges from 0-100, higher scores indicate more pain or disability

SECONDARY OUTCOMES:
Disabilities of the arm, shoulder, and hand | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure sports/music and work related to shoulder pain, ranges from 0-100, higher scores indicate more pain or disability
Visual analog scale | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder pain, ranges from 0-10, higher score indicate more pain
range of motion | score change from baseline to 1 week, 1 month and 3 months after treatment
  measure shoulder range of motion, higher score indicate higher range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No